CLINICAL TRIAL: NCT00901173
Title: The THINKER Study: A Pilot for a Case-Control of Esophageal Squamous Cell Carcinoma in Western Kenya
Brief Title: A Pilot for a Case-Control Study of Esophageal Squamous Cell Carcinoma in Western Kenya
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909141; 09-C-N141
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Case-Control Study; Esophageal Squamous Cell Carcinoma; Risk Factors
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

* Esophageal cancer is the sixth leading cause of cancer deaths worldwide. Two primary cell types, squamous cell carcinoma and adenocarcinoma, account for most cases. Of the two, esophageal squamous cell carcinoma (ESCC) accounts for more than 80 percent of all deaths from esophageal cancer. Many cases occur in certain areas with defined geographic boundaries, including parts of Kenya.
* Studies of ESCC in developed countries (such as the United States) suggest that heavy tobacco and alcohol use, poor diet, and low socioeconomic status are the primary risk factors. Males and African Americans are also at higher risk. However, these risk factors do not fully explain the prevalence of cases in several of the identified geographic areas.
* ESCC is the most common cancer seen at Tenwek Hospital in western Kenya, and a notable number of patients are 30 years of age or younger.

Objectives:

* To test the feasibility of a new protocol by recruiting visitors to Tenwek Hospital and volunteers from the general population for study purposes.
* To use the new protocol to obtain blood and urine samples from ESCC cases in Tenwek Hospital and from nonpatient volunteers.

Eligibility:

* Hospital patients and volunteers who live within 50 kilometers of Tenwek Hospital in western Kenya.

Design:

* All participants will complete a questionnaire and provide blood and urine samples for testing.

  * The questionnaire will include questions about individual and family medical history, living conditions, lifestyle, habits, and diet.
  * Blood and urine samples will be collected from all participants after the questionnaire.
* Biological samples will be shipped to the United States for further testing.
* Treatment will not be offered as part of this study.

DETAILED DESCRIPTION:
This pilot study will assess the feasibility of completing the first formal case-control study to examine etiologic factors for esophageal squamous cell carcinoma (ESCC) in Kenya and will be conducted in Western Kenya, a high-risk area for ESCC.

Esophageal cancer causes over 380,000 deaths per year and ranks as the sixth leading cause of cancer death worldwide. Two primary cell types, squamous cell carcinoma and adenocarcinoma, account for most cases. Although the rates of esophageal adenocarcinoma have risen rapidly in the United States and elsewhere, ESCC still accounts for 80% of all esophageal cancer cases in the world. Many of these cases occur in high-risk areas with sharp geographic boundaries within China, Iran, a small region of South America, South Africa, and Kenya. Studies of ESSC in economically developed countries, such as the US, point to smoking tobacco, heavy alcohol drinking, poor diets deficient in fresh fruits and vegetables, and low socioeconomic status as the main etiologic factors. Other independent risk factors may include being male and being African-American. Smoking tobacco and heavy alcohol consumption do not explain the incidence rates in the high-risk regions because these habits are less common and less intensely practiced in these high-risk areas compared to the low risk area. Also, in highrisk areas the incidence rates are similar in men and women despite differences in the rates of tobacco smoking and alcohol drinking. Therefore, it is important to consider a wide range of etiologic factors to explain the high rates of cancer in these populations.

Tenwek Hospital is a 300 bed mission hospital located in Bomet District, Rift Valley Province, approximately 200 miles from Nairobi in the west of Kenya. Tenwek serves as a primary health care facility for approximately 400,000 people, and it has become a referral center for a broader population. ESCC is the most common malignancy seen at Tenwek Hospital and the patients show a very unusual age distribution with 10% of cases less than or equal to 30 years of age.

We will conduct a pilot for a case-control study of ESCC at Tenwek Hospital, recruiting people that live within 50 km of the hospital. Initial pilot testing showed that neither hospital-visitor controls nor general-population controls were practical control sources. We now plan to test the feasibility of collecting 50 hospital-based non-cancer patient controls. We will then enroll 50 cases and 50 additional hospital-based non-cancer patient controls to test all aspects of our protocol. We will ship the biological samples collected from these individuals to the US and test their suitability for our intended assays. All subjects will be interviewed using a structured questionnaire and will be asked to provide biological samples including blood and urine. Environmental risk factors (including lifestyle, habits, and diet) will be assessed through questionnaires.

ELIGIBILITY:
* Cases:

INCLUSION CRITERIA:

1. Consent to participate in the study
2. Pathologically diagnosed with esophageal squamous cell carcinoma at Tenwek Hospital, Bomet Kenya
3. Primary residence within 50 kilometers of Tenwek Hospital, Bomet Kenya

EXCLUSION CRITERIA:

1. Does not consent to participation in the study
2. Mental impairment that precludes consenting to or completing the study questionnaire

Controls:

INCLUSION CRITERIA:

1. Consent to participation in the study
2. No previous history of malignancy
3. Primary residence within 50 kilometers of Tenwek Hospital, Bomet Kenya

EXCLUSION CRITERIA:

1. Does not consent to participation in the study
2. Mental impairment that precludes consenting to or completing the study questionnaire

Ages: 7 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ESCC patients and controls that live within 50 km of Tenwek Hospital
Sampling Method: Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Esophageal squamous cell carcinoma | At diagnosis
  determined by pathology results from endoscopic biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Christian Abnet, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Tenwek Hospital, Bornet, Kenya

REFERENCES:
- [Background] Dawsey SP, Tonui S, Parker RK, Fitzwater JW, Dawsey SM, White RE, Abnet CC. Esophageal cancer in young people: a case series of 109 cases and review of the literature. PLoS One. 2010 Nov 22;5(11):e14080. doi: 10.1371/journal.pone.0014080. PMID 21124934
- [Background] White RE, Abnet CC, Mungatana CK, Dawsey SM. Oesophageal cancer: a common malignancy in young people of Bomet District, Kenya. Lancet. 2002 Aug 10;360(9331):462-3. doi: 10.1016/S0140-6736(02)09639-3. PMID 12241722
- [Background] Nieminen MT, Novak-Frazer L, Collins R, Dawsey SP, Dawsey SM, Abnet CC, White RE, Freedman ND, Mwachiro M, Bowyer P, Salaspuro M, Rautemaa R. Alcohol and acetaldehyde in African fermented milk mursik--a possible etiologic factor for high incidence of esophageal cancer in western Kenya. Cancer Epidemiol Biomarkers Prev. 2013 Jan;22(1):69-75. doi: 10.1158/1055-9965.EPI-12-0908. Epub 2012 Nov 15. PMID 23155139